CLINICAL TRIAL: NCT03911596
Title: Cyber Physical System for Smart Corrective Eyeglasses
Brief Title: Smart Autofocusing Eyeglasses
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB # 114415; 5U01EB023048 (NIH)
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2022-11

CONDITIONS: Presbyopia
Keywords: Presbyopia, accommodation, smart eyeglasses
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Smart Autofocusing Eyeglasses — The smart eyeglasses system is meant to be a next generation alternative technology which replaces the generic eyeglasses used for correction of refractory defects in human vision. These smart eyeglasses do not fix any internal eye problems. They just externally compensate for the loss of eye focusing functions caused by presbyopia. This system is a medical assistive device which is meant to improve the quality of life of presbyopic patients.

SUMMARY:
A high-performance smart eyeglasses system with integrated sensing, actuation, control and data collection is being developed at the University of Utah. These smart eyeglasses use tunable lenses and integrated sensor technologies to correct blurred vision caused due to a major age-related condition called presbyopia.The objective of this study is to test this smart system on patients suffering from presbyopia aged 45 and above. The researchers intend to study the effect of these smart eyeglasses by qualitatively investigating the patient's visual acuity with this smart system. The results of this study and subsequent research have the potential to lead to major lifestyle improvements and better treatment for millions of presbyopic patients that are constrained by the limitation of current corrective eyeglass technologies. There are two main sources of fairly well understood problems that lead to presbyopia and loss of the eye focusing function. The adaptive eyeglasses used in these tests do not fix any of the internal eye problems. They just compensate externally for the loss of the eye focusing function caused by presbyopia. As such, the investigators intend to evaluate our system's effectiveness in terms of the sharpness of the perceived images.

DETAILED DESCRIPTION:
Eye defects occur when the eye cannot focus images from the outside world. This results in blurred vision, which sometimes is so severe that it causes visual impairment. Among the many vision defects, presbyopia is an inevitable, irreversible, universal age-related condition where the crystalline lens in the eye loses its accomodation orthe ability to change the optical power. This defect occurs as a natural result of aging and will ultimately affect any person reaching advanced enough age. It was estimated in 2005 that over 1 billion people worldwide suffered from presbyopia, with approximately 400 million suffering from near vision loss due to the lack of correction technologies.

The most inexpensive and commonly used tools to correct vision errors are fixed power eyeglasses, which haven't seen any improvement since the mid-1800s. Conventional eyeglasses are an ancient piece of technology which originated in Europe's middle ages. A major drawback of such eyeglasses is that they can only correct the lack of accomodation at a particular object distance, since they use fixed power lenses. As a result, conventional eyeglasses can produce sharp images for objects located either far away or near the observer but not both. Bifocal, multifocal and progressive lenses can partially alleviate vision defects, but at the expense of reduced and fragmented field of view. As an example, multifocal lenses have different lens powers in different regions of the lens. With such lenses, it is not possible to see objects clearly over the entire visual field. Further, the effectiveness of conventional eyeglasses is not monitored outside the optometrist's office.

The proposed smart eyeglasses system uses a combination of large-aperture fluidic lenses, ultra-light actuators, object distance sensors and embedded control, communications and computing electronics to continuously produce sharp and focused images at any object range. They can also collect the behaviour and characteristics of the observer's eyes to gauge the effectiveness of the technology and adapt to observer's visual degradation over age.

ELIGIBILITY:
Inclusion Criteria:

* Presbyopic
* Less than 1.0 diopter astigmatism
* Eyeglass prescription between -2.5 and +2.5, correctable to 20/20

Exclusion Criteria:

* Artificial intraocular lens
* Any ocular pathology that would inhibit accommodation of the natural lens

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual above 45 years of age with symptoms of presbyopia.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Accommodation response of the natural lens of the eye with smart eyeglasses technology | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Carlos H Mastrangelo, PhD, Principal Investigator — University of Utah
Locations (1):
- Moran Eye Center, University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hasan N, Banerjee A, Kim H, Mastrangelo CH. Tunable-focus lens for adaptive eyeglasses. Opt Express. 2017 Jan 23;25(2):1221-1233. doi: 10.1364/OE.25.001221. PMID 28158006
- [Background] Hasan N, Karkhanis M, Ghosh C, Khan F, Ghosh T, Kim H, Mastrangelo CH. Lightweight Smart Autofocusing Eyeglasses. Proc SPIE Int Soc Opt Eng. 2018 Jan-Feb;10545:1054507. doi: 10.1117/12.2300737. Epub 2018 Feb 22. PMID 32773917
- [Background] N. Hasan, M. Karkhanis, F. Khan, T. Ghosh, H. Kim, and C. H. Mastrangelo. Adaptive Optics for Autofocusing Eyeglasses. Imaging and Applied Optics 2017 (3D, AIO, COSI, IS, MATH, pcAOP), OSA Technical Digest (online) (Optical Society of America, 2017), paper AM3A.1.